CLINICAL TRIAL: NCT02171559
Title: Relative Bioavailability and Pharmacodynamics of Dabigatran After a Single Dose of 220 mg Dabigatran Etexilate and After 40 mg Enoxaparin s.c. for 3 Days Followed by a Single Dose of 220 mg Dabigatran Etexilate in Healthy Male and Female Volunteers (an Open-label, Randomised, Single and Multiple Dose, Two Way Crossover Phase I Study)
Brief Title: Relative Bioavailability and Pharmacodynamics of Dabigatran With Enoxaparin in Healthy Male and Female Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 1160.78
Record Dates: First submitted 2014-06-20; First posted 2014-06-24 (Estimated); Last update posted 2014-06-24 (Estimated); Status verified 2014-06

CONDITIONS: Healthy
MeSH Terms: interventions — Dabigatran

ARMS (2):
- Dabigatran etexilate capsules after enoxaparin ampoules (Experimental)
  Interventions: Drug: Enoxaparin prefilled syringes; Drug: Dabigatran etexilate capsules
- Dabigatran etexilate capsules without enoxaparin (Active Comparator)
  Interventions: Drug: Dabigatran etexilate capsules

INTERVENTIONS:
Drug: Enoxaparin prefilled syringes
  Arms: Dabigatran etexilate capsules after enoxaparin ampoules
Drug: Dabigatran etexilate capsules

SUMMARY:
To investigate the relative bioavailability and the pharmacodynamics of dabigatran after switching from enoxaparin to dabigatran etexilate as compared to dabigatran etexilate alone

ELIGIBILITY:
Inclusion Criteria:

1. Subjects were healthy males and females based upon a complete medical history, including a physical examination, vital signs (blood pressure, pulse rate), 12-lead ECG, and clinical laboratory tests
2. Age ≥18 to ≤55 years
3. Body mass index (BMI) ≥18.5 to ≤29.9 kg/m2
4. Signed and dated written informed consent prior to admission to the study in accordance with GCP and the local legislation

Exclusion Criteria:

1. Gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological, or hormonal disorders
2. Relevant surgery of gastrointestinal tract
3. History of any bleeding disorder or acute blood coagulation defect
4. Diseases of the central nervous system (such as epilepsy) or psychiatric disorders or neurological disorders
5. History of relevant orthostatic hypotension, fainting spells or blackouts
6. Chronic or relevant acute infections
7. History of allergy/hypersensitivity (including drug allergy) which was deemed relevant to the trial as judged by the investigator
8. Intake of any medication within 2 weeks of first dosing, especially intake of medication, which influences blood clotting, i.e. acetylsalicylic acid, cumarin etc.
9. Use of drugs which might reasonably influence the results of the trial based on the knowledge at the time of protocol preparation within 4 weeks prior to administration or during the trial
10. Alcohol abuse (more than 60 g/day for males and more than 20 g/day for females)
11. Drug abuse
12. Intake of grapefruit, grapefruit juice, or products containing grapefruit juice, Seville oranges, garlic supplements, or St. John's wort within 5 days of first dosing
13. Participation in another trial with an investigational drug within 2 months prior to trial drug administration or during the trial
14. Blood donation (more than 100 mL within 4 weeks prior to trial drug administration or during the trial)
15. Excessive physical activities (within 1 week prior to trial drug administration or during the trial)
16. Any laboratory value outside the reference range that was of clinical relevance
17. Inability to comply with dietary regimen of study centre
18. Smoker (>10 cigarettes or >3 cigars or >3 pipes/day)
19. Inability to refrain from smoking on trial days

    For female subjects:
20. Pregnancy / positive pregnancy test, or planning to become pregnant during the study or within 1 month after study completion
21. No adequate contraception during the study and within 1 month after study completion such as implants, injectables, combined oral contraceptives, intrauterine device, sexual abstinence (for at least 1 month prior to enrolment), vasectomised partner (vasectomy performed at least 1 year prior to enrolment), or surgical sterilisation (including hysterectomy). Females, who did not have a vasectomised partner, were not sexually abstinent or surgically sterile, were asked to additionally use a barrier contraception method (e.g. condom, diaphragm with spermicide)
22. Lactation period

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 29 (Actual)
Dates: Start 2008-08; Primary Completion 2008-09 (Actual)

PRIMARY OUTCOMES:
Area under the concentration-time curve of the analyte in plasma over the time interval from 0 extrapolated to infinity (AUC0-∞) of dabigatran | Up to 48 hours after drug administration
Maximum measured concentration of the analyte in plasma (Cmax ) of dabigatran | Up to 48 hours after drug administration
Area under the effect-time curve of the analyte in plasma over the time interval from 0 to 48 h after administration (AUEC0-48) after dabigatran alone and after dabigatran following enoxaparin administration | Up to 48 hours after drug administration
Maximum effect ratio to baseline (ERmax) after dabigatran alone and after dabigatran following enoxaparin administration | Baseline and up to 48 hours after drug administration

SECONDARY OUTCOMES:
Area under the concentration-time curve of the analyte in plasma over the time interval from 0 to the last quantifiable data point (AUC0-tz) of dabigatran | Up to 48 hours after drug administration
Time from dosing to the maximum concentration of the analyte in plasma (tmax) of dabigatran | Up to 48 hours after drug administration
Terminal rate constant in plasma (λz) of dabigatran | Up to 48 hours after drug administration
Terminal half-life of the analyte in plasma (t1/2) of dabigatran | Up to 48 hours after drug administration
Mean residence time of the analyte in the body after oral administration (MRTpo) of dabigatran | Up to 48 hours after drug administration
Apparent clearance of the analyte in plasma after extravascular administration (CL/F) of dabigatran | Up to 48 hours after drug administration
Apparent volume of distribution during the terminal phase λz following an extravascular administration (Vz/F) of dabigatran | Up to 48 hours after drug administration
Anti-FIIa activity for Dabigatran etexilate | Up to 48 hours after drug administration
Anti-FXa/anti-FIIa activity for Enoxaparin | Up to 48 hours after drug administration
Activated partial thromboplastin time (aPTT) for Dabigatran etexilate | Up to 48 hours after drug administration
Ecarin clotting time (ECT) for Dabigatran etexilate | Up to 48 hours after drug administration
Thrombin time (TT) for Dabigatran etexilate | Up to 48 hours after drug administration
Change in vital signs (blood pressure, pulse rate) | up to day 61
Change in 12-lead electrocardiogram (ECG) | up to day 61
Change in clinical laboratory tests | up to day 61
Occurrence of adverse events | Up to day 61
Assessment of global tolerability by investigator on a four point scale (good, satisfactory, not satisfactory, bad) | Day 61
Assessment of local tolerability by investigator on a four point scale (good, satisfactory, not satisfactory, bad) | day 3 of enoxaparin administration